CLINICAL TRIAL: NCT02975635
Title: Patients' Preferences for Repair Versus Replacement Restorations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Göttingen (Other)
Collaborators: Georg-Elias-Mueller-Institute of Psychology, University Goettingen (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, Dr. med. dent., Dr. rer. medic., Dr. med. dent., University Medical Center Goettingen
Other Study IDs: Repair-Patients
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Patient Preference
Keywords: Patients' Preferences
MeSH Terms: conditions — Patient Preference | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral patient information only: Patients are given oral information only (information as usual). After patients have made their decisions (repair or replacement), a questionnaire survey is conducted.
  Interventions: Other: Questionnaire
- Written patient education before oral patient information: Patients are given a flow chart in advance of oral information. After patients have made their decisions (repair or replacement), a questionnaire survey is conducted.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients are given a questionnaire with items related to personality and behaviour.

SUMMARY:
Partially defective dental restorations might either be treated by complete replacement or by repair of the affected region. Repair restorations are a scientifically proven approach to manage failed restorations, but probably unknown to most patients. Results from this study and findings on the predictors of patients' therapy decisions might improve future patient information documents.

DETAILED DESCRIPTION:
Handling insufficient restorations contributes up to 2/3 of all treatments in dentistry. Formerly, defective restorations were completely removed and replaced. Today, repair restorations are an alternative choice. During repair treatment, only the defective portion of a restoration (instead of the complete restoration) is removed and replaced. By performing repair restorations dental hard tissue can be conserved and the risk of treatment associated complications is reduced.

Recent studies have shown that survival rates of repair restorations are slightly lower compared to replacement fillings. Nevertheless, in certain clinical situations repair restorations are more cost-effective than replacement.

Further studies have shown that patients' decisions differ with regard to a variety of factors. This applies to decisions regarding dental treatments as well. However, patients' decisions between both possible therapy options (repair or replacement) of partially defective restorations are not yet investigated.

ELIGIBILITY:
Participant are selected by consecutive patient sampling.

Inclusion Criteria:

* At least one partially defective dental restoration which can either be repaired or replaced

Exclusion Criteria:

* Non-fulfillment of the inclusion criteria
* Lack of capacity to consent
* No German language skills in written and spoken language
* Age <18 years
* Defective restoration must be completely replaced in any event or is not suitable for repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Preventive Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Completion of a questionnaire | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr. med. dent., Principal Investigator — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Locations (1):
- University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwendicke F, Mostajaboldave R, Otto I, Dorfer CE, Burkert S. Patients' preferences for selective versus complete excavation: A mixed-methods study. J Dent. 2016 Mar;46:47-53. doi: 10.1016/j.jdent.2016.01.006. Epub 2016 Jan 18. PMID 26796700
- [Background] Weeks L, Balneaves LG, Paterson C, Verhoef M. Decision-making about complementary and alternative medicine by cancer patients: integrative literature review. Open Med. 2014 Apr 15;8(2):e54-66. eCollection 2014. PMID 25009685
- [Background] Ernst J, Brahler E, Weissflog G. [Patient involvement in medical decision making--an overview on patient preferences and impacting factors]. Gesundheitswesen. 2014 Apr;76(4):187-92. doi: 10.1055/s-0033-1361150. Epub 2014 Jan 9. German. PMID 24408309
- [Background] Kanzow P, Hoffmann R, Tschammler C, Kruppa J, Rodig T, Wiegand A. Attitudes, practice, and experience of German dentists regarding repair restorations. Clin Oral Investig. 2017 May;21(4):1087-1093. doi: 10.1007/s00784-016-1859-3. Epub 2016 Jun 2. PMID 27255959
- [Background] Kanzow P, Wiegand A, Schwendicke F. Cost-effectiveness of repairing versus replacing composite or amalgam restorations. J Dent. 2016 Nov;54:41-47. doi: 10.1016/j.jdent.2016.08.008. Epub 2016 Aug 26. PMID 27575986